CLINICAL TRIAL: NCT00183833
Title: Phase I/II Study of Xeloda and Gleevec in Patients With Advanced Solid Tumors
Brief Title: Study of Xeloda and Gleevec in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3C-02-1
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Colon Cancer; Colorectal Cancer
Keywords: phase 1; phase I; phase one; colon cancer; colorectal cancer
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms | interventions — Capecitabine; Imatinib Mesylate

ARMS (1):
- A (Experimental): Xeloda plus gleevec
  Interventions: Drug: capecitabine, imatinib mesylate

INTERVENTIONS:
Drug: capecitabine, imatinib mesylate — Capecitabine and imatinib mesylate will both be taken by mouth twice a day

SUMMARY:
This study is for people with solid tumors cancer for which the standard chemotherapy drugs have not worked. The purpose of this research is to evaluate the side effects of Xeloda (also called capecitabine) in combination with a new anticancer agent called Gleevec (also called imatinib mesylate). Xeloda is an anticancer drug, and can be taken by mouth. The active ingredient is a well-studied cancer drug called 5-FU. Xeloda is approved by the FDA for the treatment of colon cancer. Gleevec is approved in the US for the treatment of patients with a leukemia called CML (increase of white blood cells) after failure of standard therapy. It is also approved by the FDA for patients with Gastrointestinal Stromal Tumors (a rare tumor in the digestive tract).

This study will test how much Gleevec we can safely give with Xeloda. Xeloda will be given at the recommended dose for colorectal cancer and Gleevec will be given in increasing amounts.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic or unresectable solid tumor for which standard curative or palliative measures do not exist or are no longer effective.
* SWOG performance status 0-2.
* ANC greater than 1500, platelets greater than 100,000.
* Total bilirubin less than 2 x upper limit of normal, or less than 3 x upper limit of normal in patients with liver metastasis. Transaminase (AST and/or ALT) less than 2 x upper limit of normal or less than 3 x upper limit of normal in patients with liver metastasis.
* Serum creatinine less than 1.25 x institutional upper limit of normal.
* Female patients of childbearing potential must have negative pregnancy test within 7 days before initiation of study drug dosing.

Exclusion Criteria:

* Patient has received any other investigational agent- within 28 days of first day of study drug dosing.
* Patient with another primary malignancy except if the other primary malignancy is neither currently clinically significant nor requiring active intervention.
* Patient has another severe and/or life-threatening medical disease.
* Patient has an acute or known chronic liver disease (e.g., chronic active hepatitis, cirrhosis).
* Patient has a known diagnosis of human immunodeficiency virus (HIV) infection.
* Patient has received chemotherapy within 4 weeks (6 weeks for nitrosourea, mitomycin-C or any antibody therapy) prior to study entry unless urgent enrollment needed and approved by Novartis.
* Patient had a major surgery within 2 weeks prior to study entry.
* Patients with symptomatic brain metastasis.
* Patient with Grade III/IV cardiac problems as defined by the New York Heart Association Criteria (e.g. congestive heart failure, myocardial infarction within 6 months of study)
* Medical, social or psychological factors interfering with compliance.
* Patients under therapeutic coumadin therapy.
* Patients under routine systemic corticosteroid therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2002-12; Primary Completion 2009-07 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
To determine the dose limiting toxicity (DLT) and maximum tolerated dose (MTD) of Gleevec in combination with a fixed dose of Xeloda po bid daily in patients with colon cancer. | 4 weeks

SECONDARY OUTCOMES:
To determine the time to progression, survival and response rate. | Until Patient goes off study
To obtain preliminary data on molecular correlates to determine clinical efficacy | Until Patient Goes off study
Toxicity. | 30 days after patient receives last drug dose

CONTACTS AND LOCATIONS:
Overall Officials: Heinz-Josef Lenz, M.D., Principal Investigator — U.S.C./Norris Cancer Center
Locations (1):
- USC/Norris Cancer Center, Los Angeles, California, United States